CLINICAL TRIAL: NCT01215305
Title: A Cross-sectional Study on the Prevalence and Extraesophageal Symptoms of GERD in Patients With Upper GI Symptoms, Visiting the Outpatient Departments of Peripheral Hospitals in Greece. The 'GERDQ-XS' Study
Brief Title: A Cross-sectional Study on the Prevalence and Extraesophageal Symptoms of Gastroesophageal Reflux Disease(GERD) in Patients With Upper GI Symptoms, Visiting the Outpatient Departments of Peripheral Hospitals in Greece
Acronym: GERDQ-XS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Panagiotis Pontikis/MC MD, AstraZeneca S.A. Greece
Other Study IDs: NIS-GGR-DUM-2010/1
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2011-04

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux Disease, extraesophageal symptoms
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Visiting outpatient departments, if symtoms: patients with upper GI symptoms, visiting the outpatient departments of peripheral hospitals in Greece

SUMMARY:
The present study has been designed to provide current data on GERD prevalence in several regional areas of Greece outside the two major urban centres (Athens and Thessaloniki), to measure the treatment response in GERD patients, and to assess the correlations between the two methods of diagnosing GERD, i.e. reporting of symptoms by the patient to the physician and completion of the GerdQ questionnaire by the patient. Additionally, this study aims to provide data on the prevalence of extraesophageal symptoms in GERD patients in Greece. The XQS questionnaire will be applied for the identification of these patients and the assessment of the extraesophageal disease burden (frequency and intensity/severity). Finally, an association between the GerdQ and XQS scores will be attempted.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Patients aged 18 and over
* Patients with upper-GI symptoms during the last week prior to the study visit

Exclusion Criteria:

* History of oesophageal, gastric or duodenal surgery
* Patients with history of malignancy
* Treatment with acetylsalicylic acid/NSAID during the last week prior to the study visit
* Therapy with PPI for the healing of ulcer induced by treatment with acetylsalicylic acid/NSAID
* Therapy with PPI for HP eradication or for healing of HP-related peptic ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with upper GI symptoms
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
GerdQ score | End of recruitment (estimated timeframe :2.5 months)

SECONDARY OUTCOMES:
Demographic data (age, gender, race, weight, height) | End of recruitment (estimated timeframe :2.5 months)
Marital status | End of recruitment (estimated timeframe :2.5 months)
Smoking habits, alcohol consumption | End of recruitment (estimated timeframe :2.5 months)
Patient's eating habits and implementation of dietary recommendations | End of recruitment (estimated timeframe :2.5 months)
Place of residence (urban, suburban, rural) | End of recruitment (estimated timeframe :2.5 months)
Education level | End of recruitment (estimated timeframe :2.5 months)
Occupation | End of recruitment (estimated timeframe :2.5 months)
General medical history | End of recruitment (estimated timeframe :2.5 months)
History of upper gastrointestinal diseases | End of recruitment (estimated timeframe :2.5 months)
Way of antisecretory treatment administration for GI symptoms the last month prior to study visit (if applicable) | End of recruitment (estimated timeframe :2.5 months)
Compliance to antisecretory treatment (if applicable) | End of recruitment (estimated timeframe :2.5 months)
Upper GI symptomatology XQS score | End of recruitment (estimated timeframe :2.5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Pontikis, Study Director — AstraZeneca
Locations (19):
- Greece (19):
  - Research Site, Chania, Crete
  - Research Site, Rhodes, Dodekanis
  - Research Site, Ioannina, Ipiros
  - Research Site, Preveza, Ipiros
  - Research Site, Áno Sýros, Kyklades
  - Research Site, Chalkidiki, Makedonia
  - Research Site, Edessa, Makedonia
  - Research Site, Kavala, Makedonia
  - Research Site, Serres, Makedonia
  - Research Site, Limnos, NE Aegian
  - Research Site, Kalamata, Peloponisos
  - Research Site, Kalávryta, Peloponisos
  - Research Site, Moláoi, Peloponisos
  - Research Site, Sparti, Peloponisos
  - Research Site, Karditsa, Thesalia
  - Research Site, Larissa, Thesalia
  - Research Site, Trikala, Thesalia
  - Research Site, Volos, Thesalia
  - Research Site, Komotini, Thraki